CLINICAL TRIAL: NCT03295045
Title: Evolution of the Profile of Infectious Endocarditis in France in 2008
Brief Title: Evolution of the Profile of Infectious Endocarditis in France in 2008 (EI2008)
Acronym: EI2008
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Bichat Hospital (Other); Hopital Louis Pradel (Other); Central Hospital, Nancy, France (Other); University Hospital, Montpellier (Other); CHU de Reims (Other); Rennes University Hospital (Other); Hotel Dieu Hospital (Other); Henri Mondor University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: N/2007/50
Record Dates: First submitted 2017-09-05; First posted 2017-09-27 (Actual); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Infective Endocarditis
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Infective endocarditis (IE) is a rare (30 cases / million / year in France) and serious (20 % of deaths during hospitalization) disease . Its epidemiological profile was considerably modified these last years.New predisposing factors appeared, due to increasing number of patients wearing valvular prosthetics. The purpose of this study is to realize in 2008 a new observational study on populational basis to describe and analyze the evolution of the epidemiology of IE in France, compared to previous studies conducted in 1991 and 1999.

DETAILED DESCRIPTION:
It is a prospective observational study based on a population of 25 million inhabitants. The cases are recruited over a one year period, from January 1st till December 31st, 2008, in six regions of France (Rhône-Alpes, Paris et Petite Couronne, Lorraine, Franche-Comté, Marne, Languedoc-Roussillon) and in the department of Ille-et-Vilaine. The IE cases are declared by clinicians taking care of the patients, microbiologists and cardiac ultrasonographists.

ELIGIBILITY:
Inclusion Criteria:

* Major Patient
* Supported in one of the participating centers
* The application of diagnostic classification criteria of Duke modified by Li is carried out after collection of all the data at the output of the patient. Will be included in the observatory that patients meeting criteria for definite or possible endocarditis.

  * Affiliated with the French social security regime

Exclusion Criteria:

* Patients not living in one of the studied regions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients with infective endocarditis living in one of the studied regions
Sampling Method: Non-Probability Sample
Enrollment: 484 (Actual)
Dates: Start 2007-12-01 (Actual); Primary Completion 2009-12-31 (Actual); Study Completion 2010-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | 1 year
  Vital status

SECONDARY OUTCOMES:
Frequency of antibiotic resistance by the germs (streptococci and staphylococci) | during the hospitalization, 1 year maximum
  antibiotic treatments and outcome

CONTACTS AND LOCATIONS:
Overall Officials: Bruno HOEN, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Pointe à Pitre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Selton-Suty C, Celard M, Le Moing V, Doco-Lecompte T, Chirouze C, Iung B, Strady C, Revest M, Vandenesch F, Bouvet A, Delahaye F, Alla F, Duval X, Hoen B; AEPEI Study Group. Preeminence of Staphylococcus aureus in infective endocarditis: a 1-year population-based survey. Clin Infect Dis. 2012 May;54(9):1230-9. doi: 10.1093/cid/cis199. PMID 22492317
- [Result] Duval X, Delahaye F, Alla F, Tattevin P, Obadia JF, Le Moing V, Doco-Lecompte T, Celard M, Poyart C, Strady C, Chirouze C, Bes M, Cambau E, Iung B, Selton-Suty C, Hoen B; AEPEI Study Group. Temporal trends in infective endocarditis in the context of prophylaxis guideline modifications: three successive population-based surveys. J Am Coll Cardiol. 2012 May 29;59(22):1968-76. doi: 10.1016/j.jacc.2012.02.029. PMID 22624837